CLINICAL TRIAL: NCT05224297
Title: Patient Experience Data in Radiation Oncology
Acronym: PEDRO
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerd Heilemann, Principal Investigator, Medical University of Vienna
Other Study IDs: 2184/2019
Record Dates: First submitted 2022-01-25; First posted 2022-02-04 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Radiotherapy Side Effect; PROMs
Keywords: radiation oncology; patient reported outcome
MeSH Terms: conditions — Radiation Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (9):
- breast
  Interventions: Radiation: external beam photon therapy
- thorax
  Interventions: Radiation: external beam photon therapy
- skin
  Interventions: Radiation: external beam photon therapy
- abdomen
  Interventions: Radiation: external beam photon therapy
- skull
  Interventions: Radiation: external beam photon therapy
- head and neck
  Interventions: Radiation: external beam photon therapy
- pelvis male
  Interventions: Radiation: external beam photon therapy
- pelvis female
  Interventions: Radiation: external beam photon therapy
- extremities
  Interventions: Radiation: external beam photon therapy

INTERVENTIONS:
Radiation: external beam photon therapy — Patients receive external beam photon therapy for different tumor locations (groups).

SUMMARY:
The project is part of the overarching goal of improving patient-centric radiation oncology. This pilot project aims to develop an instrument that can be used to collect clinically relevant patient-reported outcome data on adverse effects during and after RT. This real-world evidence (RWE) database will be the basis to monitor and evaluate future technological developments, combination treatments (e.g. radioimmunotherapy, etc.), or changes in treatment protocols. The pseudonymized data will be linked to data in the oncological information system and dosimetric data from the treatment planning system. In this way, they represent a basic building block of patient-oriented development of clinical radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* all patients receiving external beam radiotherapy

Exclusion Criteria:

* unable to independently answer questionnaires on radiation-induced side effects

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is aimed to include a comprehensive representative cross-section for each of the study groups.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
radiation-related side effects | during radiotherapy and after (up until 5 years)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No